CLINICAL TRIAL: NCT00415922
Title: A Randomized, Two-Way Crossover Study to Investigate the Bioavailability of a Single Oral Dose of 37.5 mg Carbidopa, 150 mg Levodopa and 200 mg Entacapone Compared to a Single Oral Combined Dose of Both 37.5 mg Carbidopa and 150 mg Levodopa and 200 mg Entacapone in Healthy Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Carbidopa/Levodopa/Entacapone Combination vs. Carbidopa/Levodopa Combination Plus Entacapone in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CELC200A2104
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: Bioequivalence; bioavailability; carbidopa; levodopa; entacapone; fasting condition; Healthy volunteers study
MeSH Terms: interventions — Stalevo

INTERVENTIONS:
Drug: ELC200 (carbidopa+levodopa+entacapone)

SUMMARY:
The purpose of this study is assess the safety and bioequivalence of a single oral dose of carbidopa+levodopa+entacapone combination versus a single oral dose of carbidopa+levodopa combination plus a single oral dose of entacapone under fasting conditions in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects age 18 to 55 years of age included, and in good health
* At Screening, and Baseline, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed after the subject has rested for at least five (5) minutes, and again when required after three (3) minutes in the standing position. Vital signs should be within the normal ranges
* Body mass index (BMI) within the range of 18 to 27 and weigh at least 50 kg
* Female subjects must have undergone hysterectomy, or must be postmenopausal.

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin
* Receiving monoamine oxidase (MAO) inhibitors within 28 days prior to the first dose
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result
* History of clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or drugs similar to the study drug.
* Significant illness within two weeks prior to dosing
* Subjects who, through completion of the study, would have donated in excess of: 500 mL of blood in 14 days; 1500 mL of blood in 180 days; 2500 mL of blood in 1 year.
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.
* Women of child bearing potential ( WOCBP)
* History or presence of glaucoma or any suspicious undiagnosed skin lesions

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42
Dates: Start 2006-07

PRIMARY OUTCOMES:
Bioequivalence between 37.5 mg carbidopa/150 mg levodopa/200 mg entacapone single dose combination and 37.5 mg carbidopa/150 mg levodopa single dose combination plus 200 mg entacapone single dose when administered under fasting conditions

SECONDARY OUTCOMES:
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Nuremberg, Germany